CLINICAL TRIAL: NCT04259385
Title: Effects of Sugary Drink Warning Labels on Parent Choices for 6-11 Year Olds
Brief Title: Effects of Sugary Drink Warning Labels on Parent Choices
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely during COVID-19 outbreak (only 1 participant)
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Drexel University (Other); University of Connecticut (Other); New York University (Other); University of Delaware (Other)
Responsible Party: Principal Investigator, Christina Roberto, PHD, Assistant Professor of Medical Ethics & Health Policy, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01DK111558_2; R01DK111558 (NIH); 33648 (Registry Identifier: AsPredicted)
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Food Preferences
Keywords: Food labeling; Child; Sugar-sweetened beverages; Eating; Drinking; Choice behavior
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Intervention Model Description: This randomized, controlled lab-based study will capture beverage and snack purchases from a concession stand and measure how much participants consume while watching a television show. Participants will be randomized to 1 of 3 groups: 1) calorie labels (control); 2) text warning labels; or 3) graphic warning labels displaying amounts of sugar.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Calorie/Control Label Condition (Active Comparator): Beverages at the concession stand and in the parent survey in this arm will display solely a calorie label.
  Interventions: Behavioral: Exposure to beverage calorie information
- Text Warning Label Condition (Experimental): Sugary beverages at the concession stand and in the parent survey in this arm will display both a text warning and a calorie label.
  Interventions: Behavioral: Exposure to sugar-sweetened beverage warning labels; Behavioral: Exposure to beverage calorie information
- Sugar Graphic Label Condition (Experimental): Sugary beverages at the concession stand and in the parent survey in this arm will display a sugar graphic warning label depicting the amount of sugar in the product, the same text warning, and a calorie label.
  Interventions: Behavioral: Exposure to sugar-sweetened beverage warning labels; Behavioral: Exposure to beverage calorie information

INTERVENTIONS:
Behavioral: Exposure to sugar-sweetened beverage warning labels — Graphic images of the amount of sugar (randomly assigned teaspoons, packets, or cubes) and text warning labels
  Arms: Sugar Graphic Label Condition; Text Warning Label Condition
Behavioral: Exposure to beverage calorie information — Calories for sugar-sweetened and non-sugar-sweetened beverages

SUMMARY:
Sugar-sweetened beverages (SSBs) are a significant contributor to adult and childhood obesity. Policies to place health warning labels on sugar-sweetened beverages are being pursued, but there is little empirical data on how such labels influence people. The proposed research will evaluate the impact of different types of sugar-sweetened beverage warning labels relative to standard calorie labels on the purchasing and consumption behaviors of parents and children.

DETAILED DESCRIPTION:
The primary objective of this proposal is to determine, before wide-scale implementation, to what degree SSB warning labels increase consumers' knowledge about the potential health harms of SSBs and reduce SSB intake. The study is designed to answer two additional questions: 1) Do some warning labels work better than others? 3) If warning labels influence behavior, is it because they increase knowledge or simply provide a salient reminder that some drinks are less healthy? This aim is designed to test the effect of warning labels on total kilocalories (kcals) purchased and consumed by parents and children. We will examine how SSB warning labels influence snack and beverage purchases and intake among 405 racially and ethnically diverse parent-child pairs.

ELIGIBILITY:
Inclusion Criteria:

* Participant pairs must be:
* Primary caregiver of a child 6-11 years old; 18 years or older; can read and speak English; did not participate in related studies from our group
* Child is between 6 and 11 years old; drinks SSBs at least 12 times per month (~3 times per week)

Exclusion Criteria:

* Unable to participate in person in Philadelphia
* Parent did not purchase food and beverage for their child
* Parent or caregiver refused to give child permission to participate

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Total beverage calories purchased for the child | Study visit, one hour
  Total number of calories for all beverages purchased for the child during the study visit
Total calories purchased for the child | Study visit, one hour
  Total number of calories for all food and beverages (summed) purchased for the child during the study visit
Total calories the child consumes | Study visit, one hour
  Total number of calories consumed by the child for all food and beverages (summed) during the study visit

SECONDARY OUTCOMES:
Total beverage calories purchased for the adult | Study visit, one hour
  Total number of calories for all beverages purchased for the adult during the study visit
Total calories purchased for the adult | Study visit, one hour
  Total number of calories for all food and beverages (summed) purchased for the adult during the study visit
Beverage calories the child consumes | Study visit, one hour
  Total number of calories consumed by the child for all beverages during the study visit
Beverage calories the adult consumes | Study visit, one hour
  Total number of calories consumed by the adult for all beverages during the study visit
Total calories the adult consumes | Study visit, one hour
  Total number of calories consumed by the adult for all food and beverages (summed) during the study visit

OTHER OUTCOMES:
Parent sugary beverage purchase intentions for the child | Study visit, 1 hour
  Average of intentions for 4 sugary beverages (1 (not at all likely) - 5 (extremely likely))
Parent non-sugary beverage purchase intentions for the child | Study visit, 1 hour
  Average of intentions for 3 non-sugary beverages (1 (not at all likely) - 5 (extremely likely))
Sugary beverage health beliefs and risk perceptions for the child | Study visit, 1 hour
  Average of 9 summed items for 4 sugary beverages (1 (strongly disagree) - 5 (strongly agree))
Non-sugary beverage health beliefs and risk perceptions for the child | Study visit, 1 hour
  Average of 9 summed items for 3 non-sugary beverages (1 (strongly disagree) - 5 (agree))
Sugary beverage accuracy of calorie knowledge | Study visit, 1 hour
  Average of difference between actual calories in each item from the calories reported by participants across 4 sugary beverages (larger numbers = overestimation)
Non-sugary beverage accuracy of calorie knowledge | Study visit, 1 hour
  Average of difference between actual calories in each item from the calories reported by participants across 3 non-sugary beverages (larger numbers = overestimation)
Sugary beverage accuracy of sugar knowledge | Study visit, 1 hour
  Average of difference between actual teaspoons of sugar in each item from the number of teaspoons reported by participants across 4 sugary beverages (larger numbers = overestimation)
Non-sugary beverage accuracy of sugar knowledge | Study visit, 1 hour
  Average of difference between actual teaspoons of sugar in each item from the number of teaspoons reported by participants across 3 non-sugary beverages (larger numbers = overestimation)
Sugary beverage categorical perception of amount of sugar | Study visit, 1 hour
  Proportion of 4 sugary beverages coded as just right or too much vs. none or too little
Non-sugary beverage categorical perception of amount of sugar | Study visit, 1 hour
  Proportion of 3 non-sugary beverages coded as none vs. all other options

CONTACTS AND LOCATIONS:
Overall Officials: Christina A Roberto, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No